CLINICAL TRIAL: NCT03633279
Title: Treatment of Sarcopenia Improves the Muscle Mass and Muscle Strength of Patients With Liver Cirrhosis- Child C: A Randomized Double Blind Control Trial
Brief Title: Treatment of Sarcopenia Improves the Muscle Mass and Muscle Strength of Patients With Liver Cirrhosis-Child C
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dayanand Medical College and Hospital (Other)
Responsible Party: Principal Investigator, Prof. Sandeep S Sidhu, Professor, Dayanand Medical College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIMM 2018
Record Dates: First submitted 2018-06-20; First posted 2018-08-16 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-08

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Amino Acids, Branched-Chain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Branched Chain Amino Acid (Experimental): Branched Chain amino acid 10 grams packet (L-Isoleucine (952 Mg), L-Leucine (1904 Mg.), L-Valine(1144 Mg). one packet at 6pm and two at 9pm.
  Interventions: Drug: Branched chain amino acid
- Placebo (Placebo Comparator): Equinitrogenous amount of lactoalbumin 2.1 grams, and equicaloric amount with 4.0 g saccharose and 3.0 g mannitol for a total of 33.6 kcal/packet.(one packet at 6pm and two at 9pm)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Branched chain amino acid — Branched chain amino acid 10 grams packet (L-Isoleucine (952 Mg), L-Leucine (1904 Mg.), L-Valine(1144 Mg).
  Arms: Branched Chain Amino Acid
Drug: Placebo — an equinitrogenous amount of lactoalbumin 2.1 grams, and equicaloric amount with 4.0 g saccharose and 3.0 g mannitol for a total of 33.6 kcal/packet.(one packet at 6pm and two at 9pm)
  Arms: Placebo

SUMMARY:
Sarcopenia is defined as loss of skeletal muscle mass. In cirrhosis, due to impaired urea genesis and decreased hepatic ammonia disposal, the skeletal muscle functions as a metabolic partner for the liver. The proportion of patients with sarcopenia is higher in those with alcoholic liver cirrhosis (80%) compared to cirrhosis due to other etiologies (31%-71%).

Sarcopenia is prevalent in > 50% patients with Child C cirrhosis. Sarcopenia increases the risk for severe infections in patients with cirrhosis. Adequate amino acid supply is needed for appropriate antibody and cytokine responses, that is impaired when skeletal muscle mass. The sepsis-related mortality rates in patients with and without sarcopenia are 22% and 8%, respectively (P = 0.02). In patients with liver cirrhosis is protein-calorie malnutrition, leading to severe consequences to the general state and clinical evolution of the patient.

DETAILED DESCRIPTION:
Globally, the mortality after any infection in cirrhosis patients is very high. The cumulative mortality in patients with infections was 43.5% (11,987 patients) where as the mortality rate without infection was 13.6% (2317 patients). Over the years, variceal bleeding causing death in cirrhosis has declined substantially but there has been no improvement in infection causing mortality over several decades. It adversely affects clinical outcomes including survival, quality of life, development of other complications.

Radiological image analysis is currently used to diagnose sarcopenia in cirrhosis. The European Working Group on Sarcopenia in Older People and Wilson D et al, recommend using the presence of both low muscle mass and low muscle function (strength or performance) for the diagnosis of sarcopenia.

Cirrhosis is believed to be a state of anabolic resistance and standard replacement of nutrients are generally ineffective.

Patients with cirrhosis frequently show protein and energy deficiency. Protein deficiency leads to hypoalbuminemia, inducing ascites and edema, whereas energy deficiency decreases fat and muscle mass and causes muscle weakness, decreasing the quality of life of patients with cirrhosis. Moreover, in patients with advanced chronic liver disease, Branched Chain Amino acids concentrations are low, whereas the concentrations of aromatic amino acids such as phenylalanine and tyrosine are high, conditions that may be closely associated with hepatic encephalopathy and the prognosis of these patients. The survival rate of patients with sarcopenia liver cirrhosis has been found to be significantly lower than that of non-sarcopenia cirrhotic patients. Long-term Branched Chain Amino acids supplementation significantly raises the survival rate in sarcopenia liver cirrhosis but not in non-sarcopenia liver cirrhosis showed that sarcopenia was associated with mortality in patients undergoing Live Donor Liver Transplantation, and perioperative nutritional therapy significantly improved overall survival in patients with sarcopenia.

It has been reported that the longer the duration on a waiting list for liver transplantation, the more sarcopenia the patient has become, even though their Model for End-stage Liver Disease scores stay the same. Patients in an advanced state of sarcopenia are confronted by their vulnerability to infection, and ultimately their imminent death. Patients with sarcopenia tended to have postoperative complications, especially infectious complications. Studies differ on the effect of of Sarcopenia on post transplant mortality. Montano-Loza et al reported that patients with "extreme" sarcopenia exhibited significantly worse prognosis. Nevertheless, patients with severe sarcopenia must have worse prognoses because of the vulnerability to infectious problems.

The main immunosuppressants used in liver transplant recipients are calcineurin inhibitors. Although liver transplant recipients usually gain weight after transplantation, that gain is mainly caused by the accumulation of fat, while skeletal muscle mass rather decreases. The state of sarcopenia rather worsen after liver transplantation. reported that sarcopenia continued to be a risk factor for mortality even in patients who managed to survive their early post transplant periods. Because sarcopenia continues, or rather worsens in some recipients, after liver transplantation, their vulnerability to infections, frailty syndrome in general, caused by sarcopenia should be seriously cautioned in addition to the problems relating to immunosuppressants.

With regard to nutritional intervention for sarcopenia, Branched Chain Amino acids supplementation is vital because Branched Chain Amino acids are an essential amino acid substrate for protein synthesis and energy generation in skeletal muscles. Branched Chain Amino acids are a group of three essential amino acids comprising valine, leucine and isoleucine; these account for 35% of the essential amino acids in skeletal muscle proteins. In patients with liver cirrhosis, Branched Chain Amino acids is not only a substrate of protein synthesis and ammonia detoxification, but is also a source of energy for the skeletal muscles.

Therefore, the consumption of Branched Chain Amino acids by skeletal muscle is accelerated in Liver Cirrhosis, leading to muscle protein breakdown, and resulting in sarcopenia As an effect on cirrhotic patients, Branched Chain Amino acids supplementation has been demonstrated to improve Protein Energy Malnutrition, raise serum albumin levels, and subsequently improve quality of life and prognosis The possible effect of Branched Chain Amino acids on sarcopenia is that leucine primarily activates the mammalian target of rapamycin signaling pathway involved in muscle protein synthesis, and additionally stimulates the pancreatic β cells to release insulin, which has an anabolic effect in skeletal muscle.

The present study demonstrated that Branched Chain Amino acids supplementation significantly improves the prognosis of sarcopenia liver cirrhosis, but its direct effect on sarcopenia itself remains unknown.

Several clinical trials have suggested that Branched Chain Amino acids supplementation improves the prognosis of cirrhotic patients. For example, a multicenter randomized trial from Italy showed that oral Branched Chain Amino acids supplementation in patients with advanced cirrhosis prevented progressive hepatic failure and improved surrogate markers and perceived health status.

The standard of care for nutrition in patients with liver cirrhosis are as follows - Nutritional recommendations target the optimal supply of adequate substrates related to requirements linked to energy, protein, carbohydrates, lipids, vitamins and minerals.

Based on these basic observations, patients with advanced chronic liver disease have been treated clinically with Branched Chain Amino acids-rich medicines, with positive effects.

Branched Chain Amino acids will complement frequent feeding with late evening snacks in reversing muscle loss in cirrhosis. The diet combined with resistance exercises shall increase skeletal muscle mass.

Clinical and laboratory Assessment Complete medical record regarding the cirrhosis, its aetiology, complications and co-morbidities will be noted. Liver Function test, Renal function test, Prothrombin time/international normalized ratio will be recorded. The severity of cirrhosis will be assessed using the Child- Pugh score and the Model of End Stage Liver Disease score.

Testing- Assessment of sarcopenia

Patients will participate in the following 4 procedures to measure sarcopenia:

1. L3 Skeletal Muscle Index Skeletal muscle area derived from a single slice CT has become more easily reproducible, and reduces the radiation exposure required to only 2.6 millisieverts. Measuring cross-sectional muscle area at either the level of the third (L3) or fourth (L4) lumbar vertebrae has been shown to correlate well with total body muscle mass (r = 0.71). When adjusted for patient height to take stature into account it is referred to as skeletal muscle index. Skeletal muscle index will be calculated from Slice-O-matic software, version 5 (Tomovision), Montreal, QC, Canada). Skeletal muscle index has been shown to be of higher accuracy in the diagnosis of sarcopenia in cirrhosis than anthropometry or dual-energy x-ray absorptiometry (DEXA) scanning and is now the most commonly employed method in studies investigating sarcopenia in cirrhosis. Diagnostic criteria have been extrapolated from Western cirrhosis populations. Multiple studies in cirrhosis, which have employed this definition, have produced clinically meaningful results and it is increasingly accepted as the most appropriate definition of sarcopenia when using cross-sectional imaging.
2. Muscle strength:It is assessed by grip strength and measured using a Jamar dynamometer. The summary of measures are as follow.

   Posture Subject seated Arm position Shoulders adducted and neutrally rotated, elbow flexed at 90°, forearm in neutral Wrist position Wrist between 0 and 30° of dorsiflexion
3. The participant will be allowed to perform one test trial. After this, three trials followed and the best score was used for analysis. Handgrip strength will be expressed in kilogram's (Kg). Three trials for each hand will be carried out and the highest value for diagnosing sarcopenia.

3. Muscle Performance [Gait Speed Test (4-metre)]:

The test can be performed with any patient able to walk 4 meters using the instructions below:

1. Instruct the patient to walk at their normal pace. Patients may use an assistive device, if needed.
2. Ask the patient to walk down a hallway through a 1-metre zone for acceleration, a central 4-metre "testing" zone, and a 1-metre zone for deceleration (the patient should not start to slow down before the 4-metre mark).
3. Start the timer with the first footfall after the 0-metre line of the testing zone
4. Stop the timer with the first footfall after the 4-metre line of the testing zone

SCORING: Gait speed of longer than 5 seconds to walk 4 meters (<0.8 m/s) suggests an increased risk of poor muscle performance.

4. Muscle Performance-The chair stand test is a physical performance test used to assess lower-extremity function. A 5 repetition test is a measure of strength; a 10 repetition test is a measure of strength and endurance. Equipment/Set Up Use a standard chair with arms and with a seat height of approximately 17 inches for all assessments, regardless of the height of the subject. Place the back of the chair against a wall to prevent movement during the test. Procedure Instruct and demonstrate the following protocol before asking the subject to perform the test:

* Sit as far back as possible in the chair seat. Keep feet firmly planted on the floor approximately hip width apart and the back of lower legs away from the chair. Keep knees bent at a 90-degree angle with arms crossed over the chest. (An individual of average or taller height will be able to sit with their upper back against the back of the chair. Individuals of shorter than average height will not be able to touch the chair back while maintaining proper position and are not required to touch the chair back during testing).
* Stand up one time and sit down, returning completely to the correct starting position.
* Indicate that any chair stands done with improper technique, e.g. not standing all the way up, not sitting all the way back, lifting feet off the floor, etc. will not be counted.
* Allow the participant the opportunity to try one chair stand to be sure when they stand up the back of their legs are not touching the chair.
* Instruct the subject that the timed assessment will begin on the command, "Ready, Set, Go" and that they are to stand up and sit back down 5 times as quickly and safely as possible. At the command "Ready, Set, Go" the tester begins timing by starting the stopwatch.
* Count each chair stand out loud when the subject is in the standing position. Provide continuous verbal encouragement during the test.
* At the tenth repetition click the stopwatch off while participant is in the standing position.
* Conduct two trials, separated by three minutes. If subjects are unable to stand up one time without assistance than they can use their hands to assist them in rising and returning to the seated position while following all other procedures as described above. Make sure to note that hands were used when recording the assessment data.

Normative value of Sarcopenia indices and association of Sarcopenia indices and mortality in child C cirrhosis patients will be also calculated.

Follow up Three months after randomization, data will be collected on the 4 objective indices of sarcopenia, as outlined above.In addition, event free survival, number of hospitalisations, combined liver events (variceal bleeds, ascites , Hepato-renal syndrome, Overt Hepatic encephalopathy, Septic complications - Pneumonias, Urinary Tract Infection, spontaneous bacterial peritonitis, skin infections and septic shock) and Quality of Life (assessed using SF 36 questionnaire) will also be recorded.

Monitoring for Adverse Events:

Branched Chain Amino acids did not increase the risk of serious adverse events, but was associated with nausea and diarrhoea. Any adverse event will be recorded specifying the time of onset, the duration, the severity and the relationship to the test medication.

Sample size: The primary objective is to show the superiority of Branched Chain Amino acids (experimental arm) versus placebo to improve both the muscle mass and muscle strength (co-primary endpoint) after 3 month of treatment in patients with sarcopeniacirrhosis (Child C) treated with standard nutrition and exercises. The co-primary endpoint is the 3-month change in CT Skeletal muscle index and Hand Grip Strength (i.e difference between the baseline and 3 month values). The study success will be only declared if both primary endpoints are statistically significant in favor of the experimental arm at two-sided significant level of 0.05. The sample size will determined as the maximum value of the sample sizes separately calculated for each endpoint with a 90% power for each comparison (considering independence between the two primary outcome as conservative approach) in order to guarantee a power of 0.80 to show the treatment efficacy on both primary outcomes. As analyzing the changes or values at 3 months are equivalent since the primary analysis will be adjusted for baseline values,Investigator determined the sample size using the 3-month values for each primary endpoints obtained in a study carried out in our center. In control arm, Investigator expect a mean CT Skeletal muscle index of 45.4±5.9 at 3-months and Mean Hand Grip Strength of 33.7+9. Compared to placebo Investigator expect that Branched Chain Amino acids will be associated with an increasing in 10% in mean value of CT Skeletal muscle index (i.e. an absolute mean difference of 4.5) and with an increasing in 20% in mean value of Hand Grip Strength (i.e. an absolute mean difference of 6.7). With a two-sided test (alpha=5%, power=90%), 38 patients per arm will be required to detect the effect size on CT Skeletal muscle index (assuming a standard deviation of 5.9) and 45 per arm to detect the effect size on Hand Grip Strength (assuming a standard deviation of 9.6). Thus, a total of 90 patients will be required. To account for an anticipated attrition rate of 20%, a total of 114 patients will be included and randomized.

Statistical Analysis Plan Statistical analyses will be independently performed by the Biostatistics Department of University of Lille under the responsibility of Professor Alain Duhamel. Data will be analyzed using the SAS software (SAS Institute Inc, Cary, NC, USA) and all statistical tests will be performed with a 2-tailed alpha risk of 0.05. A detailed statistical analysis plan will be written and finalized prior to the database lock.

All analyses will be performed for all randomized patients based on their original group of randomization, regardless of the treatment they actually received, study eligibility, or compliance post randomization, according to the intention-to-treat principle. Nis planned Baseline characteristics will be described for each arm. Quantitative variables will be expressed as mean (standard deviation), median (interquartile range) and range. Qualitative variables will be expressed as frequencies and percentages. Normality of distribution will be assessed graphically and using the Shapiro-Wilk test.

Co-Primary outcome The change in CT Skeletal muscle index and Hand Grip Strength from baseline to 3 months will be estimated and compared between the 2 arms using the constrained longitudinal data analysis model that was proposed by Liang and Zeger. The constrained longitudinal data analysis model will be used for its potential advantages compared to a conventional longitudinal analysis of covariance (ANCOVA) model. In the constrained longitudinal data analysis, both the baseline and post baseline values are modeled as dependent variables using a linear mixed model (an unstructured covariance pattern model), and the true baseline means are constrained to be the same for the 2 treatment arms. Hence, the constrained longitudinal data analysis provides an adjustment for observed baseline differences in estimating treatment effects, using all available baseline and post-baseline values. The mean between-group difference (with a 95% confidence interval(CI)) in the 3-month change in CT Skeletal muscle index and Hand Grip Strength (BCAA vs. placebo) will be estimated as an effect size with the time-by-group interaction. If normality of the model residuals is not satisfied, nonparametric analysis will be used; absolute changes between baseline and 3-month visits will be calculated and compared between the 2 arms using a non-parametric analysis of covariance that is adjusted for baseline values. The efficacy of Branched chain amino acids will be declared only if the comparison in both primary outcome is significant at p<0.05 (two-sided test).

Missing values in CT Skeletal muscle index and Hand Grip Strength measures will be handled with a multiple imputation procedure. Missing data will be imputed under the missing at random assumption (whatever the reason for missing data) by using regression switching approach (a chained equation with m=20 imputations), with the predictive mean matching method for continuous variables, and logistic regression models (binary, ordinal or polynomial) for categorical variables. The imputation procedure will be performed using main baseline characteristics and allocated arm. Treatment effect estimates that are obtained from multiple imputed data sets will be combined using Rubin's rules. Sensitivity analyses will be conducted on the observed data (case-complete analysis) and in per-protocol population. The per-protocol population will include all randomised patients who remain eligible for the study and will be 80% compliant to the allocated treatment. Any patients who will withdraw from the trial or treatment or who will not receive the allocated treatment will be excluded for per-protocol population.

Secondary outcomes The same strategy employed to analyze the co-primary outcome will be used to compare the 3-month change in muscle performance (Measured by change in Chair Stand and Gait Velocity) and the 3-month change in SF 36 - patient-reported outcome.

3-month event-free survival will be estimated using Kaplan-Meier method treating death or complications of cirrhosis as a combined events. The treatment effect will be estimated by calculating Hazard ratio (HR) and its 95% CI by using a Cox proportional hazards regression model including centers as random effect (frailty model). The proportional hazards assumption will be assessed by plotting the scaled Schoenfeld residuals of treatment effect against the rank of survival time.

Adverse events will be analyzed using descriptive analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis as diagnosed by clinical, biochemical, radiological or histologic criteria Cirrhosis - Child C class (10 - 15 score)
2. L3 SMI value < 45.4
3. Hand Grip Strength < 33.67

Exclusion Criteria:

1. Patients with hepatocellular carcinoma, in hepatic coma, with acquired immunodeficiency syndrome, with renal or pancreatic insufficiency, receiving enteral nutrition or being pregnant,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Change in CT Skeletal muscle index (cm2/m2) | 3 month
  Change in CT Skeletal muscle index (cm2/m2) (i.e difference between the baseline and 3 month values)
Change in Hand Grip Strength (Kilograms) | 3 month
  3-month change in Hand Grip Strength (Kilogram) (calculated as the difference between the baseline and 3-month values obtained by Hand Grip Dynamometer)

SECONDARY OUTCOMES:
Change in muscle performance | 3 month
  3-month change in muscle performance assessed by change in Gait Velocity (m/min)
Event-free survival | 3 month
  3-month event-free survival at 3 months (events including complications of Cirrhosis i.e. Hepatic encephalopathy, Ascites and edema, Variceal Hemorrhage, Spontaneous Bacterial Peritonitis and Hepatorenal Syndrome)
Change in Quality of life: SF 36 Scale | 3 month
  Change in health related quality of life measure by Short Form Health Survey (SF 36) QUESTIONNAIRE
Change in muscle performance | 3 month
  Change in muscle performance assessed by improvement in Chair Stand.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep s Sidhu, DM, Principal Investigator — Dayanand Medical College and Hospital, Ludhiana, Punjab, India
Locations (1):
- Dayanand Medical College and Hospital, Ludhiana, Punjab, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim G, Kang SH, Kim MY, Baik SK. Prognostic value of sarcopenia in patients with liver cirrhosis: A systematic review and meta-analysis. PLoS One. 2017 Oct 24;12(10):e0186990. doi: 10.1371/journal.pone.0186990. eCollection 2017. PMID 29065187
- [Background] Kim HY, Jang JW. Sarcopenia in the prognosis of cirrhosis: Going beyond the MELD score. World J Gastroenterol. 2015 Jul 7;21(25):7637-47. doi: 10.3748/wjg.v21.i25.7637. PMID 26167066
- [Background] Wong CH, Weiss D, Sourial N, Karunananthan S, Quail JM, Wolfson C, Bergman H. Frailty and its association with disability and comorbidity in a community-dwelling sample of seniors in Montreal: a cross-sectional study. Aging Clin Exp Res. 2010 Feb;22(1):54-62. doi: 10.1007/BF03324816. Epub 2009 Nov 25. PMID 19940555
- [Background] Merli M, Lucidi C, Giannelli V, Giusto M, Riggio O, Falcone M, Ridola L, Attili AF, Venditti M. Cirrhotic patients are at risk for health care-associated bacterial infections. Clin Gastroenterol Hepatol. 2010 Nov;8(11):979-85. doi: 10.1016/j.cgh.2010.06.024. Epub 2010 Aug 12. PMID 20621200
- [Background] Roubenoff R. Sarcopenia: effects on body composition and function. J Gerontol A Biol Sci Med Sci. 2003 Nov;58(11):1012-7. doi: 10.1093/gerona/58.11.m1012. PMID 14630883
- [Background] Montano-Loza AJ, Meza-Junco J, Prado CM, Lieffers JR, Baracos VE, Bain VG, Sawyer MB. Muscle wasting is associated with mortality in patients with cirrhosis. Clin Gastroenterol Hepatol. 2012 Feb;10(2):166-73, 173.e1. doi: 10.1016/j.cgh.2011.08.028. Epub 2011 Sep 3. PMID 21893129
- [Background] Dasarathy S, Merli M. Sarcopenia from mechanism to diagnosis and treatment in liver disease. J Hepatol. 2016 Dec;65(6):1232-1244. doi: 10.1016/j.jhep.2016.07.040. Epub 2016 Aug 8. PMID 27515775
- [Background] Wilson D, Jackson T, Sapey E, Lord JM. Frailty and sarcopenia: The potential role of an aged immune system. Ageing Res Rev. 2017 Jul;36:1-10. doi: 10.1016/j.arr.2017.01.006. Epub 2017 Feb 20. PMID 28223244